CLINICAL TRIAL: NCT05009004
Title: Digital Health for Medication Adherence Among African Americans With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Weitzman, Senior Scientist, Environment and Health Group, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R43MD015969-01A1 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: medication adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Feasibility study involving pre-post evaluation of a digital health intervention on hypertension medication adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital health intervention using text messages to support medication adherence (Experimental): In this one-arm, pre-post evaluation, all participants will receive the digital health intervention consisting of daily text messages to support medication adherence.
  Interventions: Behavioral: text messages to support medication adherence

INTERVENTIONS:
Behavioral: text messages to support medication adherence — text messages to support medication adherence

SUMMARY:
The proposed Phase 1 project aims to develop and test Memento.HTN, an individually-tailored, culturally sensitive digital health intervention comprised of a provider platform and linked patient SMS (short message service) text system to promote medication adherence among African Americans with hypertension (HTN), a group that suffers from disproportionate HTN morbidity and mortality. Memento.HTN overcomes access barriers on the part of patients and adherence support implementation barriers on the part of healthcare teams and systems. Memento.HTN is innovative in three key ways: 1) it is the first-ever linked digital provider platform and patient SMS text system for HTN medication adherence; 2) it is culturally-tailored for African Americans with HTN; and 3) it has unique monitoring functionality allowing providers to monitor individual patient adherence, support 'new start' patients, and track group adherence rates by drug class, pill format, and patient demographics.

DETAILED DESCRIPTION:
Abstract: Under the leadership of Patricia Weitzman, PhD, a multicultural, multidisciplinary team of clinicians and researchers will collaborate to develop, formatively test, and evaluate the short-effectiveness of a digital provider platform, called Memento.HTN, that is integrated with a patient SMS text system, and designed to support medication adherence by African Americans with hypertension (HTN). HTN is more common and more destructive for African Americans than for any other ethnic group. More than half of African American adults, about 15 million people, have HTN. Furthermore, African Americans are 4 times less likely to adhere to HTN medications compared to their white counterparts. Tailored approaches to reduce the racial gap in HTN morbidity and mortality, particularly those that support medication adherence, are needed in primary care. Such approaches must overcome barriers due to cost or geographic distance that can prevent African American patients from accessing adherence support. These approaches must also overcome barriers to the delivery of adherence support that stem from healthcare systems themselves. Importantly, HTN is one of most common co-morbidities in Covid19 hospitalizations, particularly for African Americans (CDC 2020).

Moreover, media coverage of a possible link between certain HTN meds, called RAAS inhibitors, and severe Covid19 outcomes may have alarmed HTN patients about the safety of their meds. As a result, the ACC (March, 2020) promptly issued guidelines recommending all patients adhere to HTN meds during the pandemic unless advised by their physicians, as there is no evidence of a link between HTN drugs and Covid19 severity. Thus, in the time of Covid19, supporting medication adherence of African Americans with HTN is extremely urgent. Memento.HTN is innovative in three key ways: 1) To our knowledge, it is the first-ever linked digital provider platform and patient SMS text system for HTN medication adherence. 2) It is culturally-tailored for African Americans with HTN. 3) It has unique monitoring functionality allowing providers to monitor individual patient adherence; support 'new start' patients, who are at increased risk for non-adherence; and track group adherence rates by drug class, pill format, and patient demographics, which have never been included in any digital med adherence intervention. Thus, the Memento.HTN system greatly simplifies and facilitates provider delivery of adherence support to patients, while enhancing their clinical therapeutics.

The provider platform sends patients interactive SMS-text pill reminders plus culturally-sensitive motivational, educational, spiritual/stress-supportive, and customizable texts, along with texts targeting intentional non-adherence and Covid19-related concerns. Texts go directly to patient cellphones (no mobile app needed), making the intervention accessible to patients who do not possess smartphones. Importantly, Memento allows 2-way texting communication between providers and patients, and automatically alerts providers when a patient has a clinically-significant pill lapse. Memento has significant commercial potential, as EHG has already developed plans for multiple digital adherence interventions that will be marketed together to clinics serving large numbers of at-risk patients. This B2B business model can generate large increases in revenues for customers, making our products attractive from both a financial and health perspective.

ELIGIBILITY:
Inclusion Criteria:

Self-identify as African American, age 18 & older, diagnosed with hypertension and on meds for it, own a cellphone (basic or smart) -

Exclusion Criteria:

Participation in other clinical research; undergoing cancer treatment; pregnancy; end stage renal disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: patricia weitzman, Principal Investigator — founder
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Health Intervention Using Text Messages to Support Medication Adherence: In this one-arm, pre-post evaluation, all participants will receive the digital health intervention consisting of daily text messages --both pill reminder text messages and motivational text messages--designed to support their daily medication adherence.
Period: Overall Study
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.36 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 22
Region of Enrollment [Number; unit: participants]
  United States | 22
Self report medication adherence [Mean (Standard Deviation); unit: units on a scale] | 87.56 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Wilson Self Report Medication Adherence Scale
Description: The self-reported medication adherence scare, developed by Wilson et al. (2016), is designed to assess self reported mediation adherence. The total scale ranges from a minimum score = 0 to a maximum score = 299.9. Higher score means better medication adherence.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
Number analyzed (Participants) | 22
units on a scale | 91.86 (9.68)

2. Primary Outcome: Hypertension Medication Adherence Self-efficacy Scale (MASES)
Description: The Hypertension MASES scale measures self efficacy for adhering hypertension medications. The scale ranges from a minimum total score = 0 to a maximum total score = 13. Higher score means greater medication adherence self efficacy.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
Number analyzed (Participants) | 22
score on a scale | 5.95 (4.66)

3. Secondary Outcome: Perceived Stress Scale
Description: The perceived stress burden scale, Cohen (1983) measures perceived stress levels. The scale ranges from a minimum total score = 0 to a maximum total score = 40. Higher total scores mean higher perceived stress.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
Number analyzed (Participants) | 22
score on a scale | 15.05 (5.20)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Digital Health Intervention Using Text Messages to Support Medication Adherence
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05009004/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05009004/SAP_001.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05009004/ICF_002.pdf